CLINICAL TRIAL: NCT01028365
Title: Time to Conceive: A Study of Fertility: Biomarkers of Fertility
Brief Title: Time to Conceive: A Study of Fertility
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R21HD060229-01A1 (NIH); UNC-Chapel Hill (Other Grant/Funding Number: 5-52208); 1R21HD060229-01A1 (NIH)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Fertility; Trying to Conceive; Trying to Get Pregnant; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Study participants will not be asked to make any changes to their daily lifestyle or existing health care routine. Participants also will not be asked to take any medications or change their diet.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Study participants will not be asked to make any changes to their daily lifestyle or existing health care routine. Participants also will not be asked to take any medications or change their diet.

SUMMARY:
The purpose of this research study is to learn a way to measure a person's fertility. After 1 year of trying, 1 out of every 7 women will not be pregnant. This is called infertility. This results in significant distress and anxiety. Infertility is common; however, the investigators have no markers to predict who will be infertile. For couples diagnosed with infertility, the investigators have used blood and urine hormone levels (follicle stimulating hormone (FSH), inhibin B, and antimullerian hormone (AMH)) to tell us who will get pregnant with fertility treatment. The investigators don't know if these hormone levels can predict if regular people trying to get pregnant will be able to get pregnant. This study will try to determine if these hormone levels can predict fertility and infertility.

ELIGIBILITY:
Inclusion Criteria:

* women between the ages of 30 and 44
* hoping to get pregnant and about to start trying or have been trying for less than 3 months
* living with male partner

Exclusion Criteria:

* currently using birth control with no intention of stopping
* have been trying to get pregnant for more than 3 months
* have used hormone shots for birth control in the past year
* have renal failure
* have known fertility problems, such as polycystic ovarian syndrome (PCOS)
* plan on moving outside of the Triangle Area in the next 6 months

Ages: 30 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women living in Chapel Hill, Raleigh, Durham, and the surrounding communities of the Triangle Area in North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2008-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Conception | 12 months, or until conception
  Examining time-to-pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Anne Z Steiner, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Su HI, Flatt SW, Natarajan L, DeMichele A, Steiner AZ. Impact of breast cancer on anti-mullerian hormone levels in young women. Breast Cancer Res Treat. 2013 Jan;137(2):571-7. doi: 10.1007/s10549-012-2361-5. Epub 2012 Dec 9. PMID 23224236
- [Background] Balthazar U, Steiner AZ. Periconceptional changes in thyroid function: a longitudinal study. Reprod Biol Endocrinol. 2012 Mar 21;10:20. doi: 10.1186/1477-7827-10-20. PMID 22436200
- [Background] Baird DD, Steiner AZ. Anti-Mullerian hormone: a potential new tool in epidemiologic studies of female fecundability. Am J Epidemiol. 2012 Feb 15;175(4):245-9. doi: 10.1093/aje/kwr439. Epub 2012 Jan 12. PMID 22247047
- [Background] Steiner AZ, Herring AH, Kesner JS, Meadows JW, Stanczyk FZ, Hoberman S, Baird DD. Antimullerian hormone as a predictor of natural fecundability in women aged 30-42 years. Obstet Gynecol. 2011 Apr;117(4):798-804. doi: 10.1097/AOG.0b013e3182116bc8. PMID 21422850
- [Result] Steiner AZ. Biomarkers of ovarian reserve as predictors of reproductive potential. Semin Reprod Med. 2013 Nov;31(6):437-42. doi: 10.1055/s-0033-1356479. Epub 2013 Oct 7. PMID 24101224
- [Result] Evans-Hoeker E, Pritchard DA, Long DL, Herring AH, Stanford JB, Steiner AZ. Cervical mucus monitoring prevalence and associated fecundability in women trying to conceive. Fertil Steril. 2013 Oct;100(4):1033-1038.e1. doi: 10.1016/j.fertnstert.2013.06.002. Epub 2013 Jul 11. PMID 23850303
- [Result] Steiner AZ, Long DL, Herring AH, Kesner JS, Meadows JW, Baird DD. Urinary follicle-stimulating hormone as a measure of natural fertility in a community cohort. Reprod Sci. 2013 May;20(5):549-56. doi: 10.1177/1933719112459226. Epub 2012 Nov 20. PMID 23171685
- [Result] Steiner AZ, Long DL, Tanner C, Herring AH. Effect of vaginal lubricants on natural fertility. Obstet Gynecol. 2012 Jul;120(1):44-51. doi: 10.1097/AOG.0b013e31825b87ae. PMID 22914390
- [Result] Mesen TB, Steiner AZ. Effect of vaginal lubricants on natural fertility. Curr Opin Obstet Gynecol. 2014 Jun;26(3):186-92. doi: 10.1097/GCO.0000000000000066. PMID 24717914
- [Derived] Crawford NM, Pritchard DA, Herring AH, Steiner AZ. Prospective evaluation of luteal phase length and natural fertility. Fertil Steril. 2017 Mar;107(3):749-755. doi: 10.1016/j.fertnstert.2016.11.022. Epub 2017 Jan 5. PMID 28065408
- [Derived] Steiner AZ, Jukic AM. Impact of female age and nulligravidity on fecundity in an older reproductive age cohort. Fertil Steril. 2016 Jun;105(6):1584-1588.e1. doi: 10.1016/j.fertnstert.2016.02.028. Epub 2016 Mar 5. PMID 26953733
- [Derived] Crawford NM, Pritchard DA, Herring AH, Steiner AZ. Prospective evaluation of the impact of intermenstrual bleeding on natural fertility. Fertil Steril. 2016 May;105(5):1294-1300. doi: 10.1016/j.fertnstert.2016.01.015. Epub 2016 Jan 25. PMID 26820771